CLINICAL TRIAL: NCT04694612
Title: Efficacy of Favipiravir in Treatment of Mild & Moderate COVID-19 Infection in Nepal: a Multi-center, Randomized, Open-labelled, Phase III Clinical Trial
Brief Title: Efficacy of Favipiravir in Treatment of Mild & Moderate COVID-19 Infection in Nepal
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nepal Health Research Council (Other Government)
Responsible Party: Principal Investigator, Dr. Prabhat Adhikari, MD, Nepal Health Research Council
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 683-2020
Record Dates: First submitted 2020-12-15; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — favipiravir; remdesivir

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomly assigned (1:1) to either Favipiravir or Placebo among mild cases; and Favipiravir or Remdesivir among moderate cases. Randomization will be stratified by age group (18 to 40 years, 40 to 60 years and 60 to 80 years) and comorbidity (presence or absence of self-reported diabetes, hypertension, Coronary Artery Disease, Coronary Heart Failure, Cancer or auto-immune disease). The permuted block (30 patients per block) randomization sequence, including stratification, will be prepared by a statistician using STATA-15 software. Once an eligible patient is enrolled in the participating center, the physician will call the central hotline that will inform the physician about the allocation based on the sequence. Eligible patients allocated to the respective arm will receive individually numbered packs, according to the sequence order as informed by the hotline.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mild condition (Placebo Comparator): Study arm groups will receive a Favipiravir treatment of 1800 mg po BID on day 1, then 800 mg po BID from day 2 onwards and control groups will receive the same quantity of Placebo.
  Duration of treatment : 5 days in each group
  Interventions: Drug: Favipiravir; Drug: Placebo
- Moderate condition (Active Comparator): Study arm groups will receive a Favipiravir treatment of 1800 mg po BID on day 1, then 800 mg po BID from day 2 onwards and control groups will receive Inj Remdesivir 200 mg IV on day 1, followed by 100 mg IV daily.
  Duration of treatment : 10 days in Favipiravir group & 5 days in Remdesivir group
  Interventions: Drug: Favipiravir; Drug: Remdesivir

INTERVENTIONS:
Drug: Favipiravir — Comparison of clinical improvement and clinical deterioration between those receiving Favipiravir compared to placebo in the patients with mild COVID-19
  Other Names: Favir 200
Drug: Placebo — Comparison of clinical improvement and clinical deterioration between those receiving Favipiravir compared to placebo in the patients with mild COVID-19
  Arms: Mild condition
Drug: Remdesivir — Comparison of clinical improvement and clinical deterioration between those receiving Favipiravir compared to Remdesivir Injection in the patients with moderate COVID-19
  Arms: Moderate condition

SUMMARY:
COVID-19 has affected almost all countries in the world. Every other country is constantly working towards its treatment and development of vaccines, with little to no success so far. Recently, several regimens have been tried as antiviral medicine. Among these medicines, Favipiravir is considered a broad-spectrum antiviral with the spectrum of activity noted against a wide range of RNA viruses & a good oral antiviral drug with > 97% bioavailability. It has already proved its safety profile as it has received FDA indication for drug-resistant Influenza. There has been increasing evidence of favorable outcome against COVID-19 in terms of early viral clearance & quicker symptomatic relief however, most of these studies lack strong statistical significance & are not peer-reviewed. Subjects will be categorized into two arms based on the severity of infection due to COVID-19 defined by NMC guidelines. Each arm will have respective two groups as the study drug group and control group. Based on the sample size calculation, subjects will be stratified & randomly enrolled in the study after checking the eligibility criteria at the screening visit. About 276 mild patients will be recruited for this trial and 400 moderate patients (including 10% loss ). Study arm groups will receive a Favipiravir treatment of 1800 mg PO BID on day 1, then 800 mg PO BID from day 2 onwards and control groups will receive the same quantity of Placebo. Treatment will be continued till 5 days after for mild groups and 10 days for moderate groups. Eligible patients will be randomly assigned (1:1) to either Favipiravir or Placebo among mild cases; and Favipiravir or Remdesivir among moderate cases. Randomization will be stratified by age group (18 to 40 years, 40 to 60 years and 60 to 80 years) and co-morbidity. The permuted block (30 patients per block) randomization sequence, including stratification, will be prepared by a statistician using STATA-15 software. Eligible patients will be allocated to the respective arm and will receive individually numbered packs, according to the sequence order as informed by the hotline. Informed written consent will be taken from the participants before commencing the study. All safety data, patient's baseline, clinical outcome data, data from endpoints and variables should be reported by the clinician and his/her team in a pre-instructed case report form (CRF) via a designated website.

It is our assumption that if the study results come favorable, Favipiravir, when used in mild or moderate cases, might prevent progression of the disease to higher severity, helps achieve viral clearance early so as to positively impact disease transmission in the community, increase the quality of life by quicker symptom recovery & decrease health burden by shortening the length of stay at the hospital. These findings can also be useful in international scenarios where the world is looking for innovative measures to curb COVID-19 infection. The study findings will be disseminated within and outside the country and will be published in peer-reviewed journals.

DETAILED DESCRIPTION:
COVID-19 stands for 2019 novel coronavirus or 2019-nCoV which is a new virus linked to the same family of viruses as Severe Acute Respiratory Syndrome (SARS), & hence named as SARS-CoV-2. It has been revealed that SARS-CoV-2 has a genome sequence that is 75%-80% identical to that of SARS-CoV. Since its first discovery in Wuhan, China in late December, it has now become a pandemic disease claiming more than nine hundred forty-five thousand deaths world-wide so far. Majority of the patients are asymptomatic or mild symptomatic, & recovery without any treatment. While there is disproportionately higher mortality among elderly & people with co-morbidities like hypertension, diabetes, obesity, heart disease or any immunocompromised status. Recently, several regimens have been tried as antiviral medicine. Among these medicines, Favipiravir is considered a broad-spectrum antiviral with spectrum of activity noted against a wide range of RNA viruses namely Influenza, West Nile virus, Yellow fever virus, Food & mouth virus, Flavivirus, Arenavirus, Bunyavirus & Alpha virus. In the USA, Japan & China, it has been approved for use in resistant Influenza. Regarding use of Favipiravir in COVID19, there have been some studies with limited data. The earlier Chinese study that compared between Favipiravir (35 patients) versus Lopinavir/Ritonavir (45 patients) among mild to moderate cases showed a trend towards earlier improvement in CT scan & quicker viral clearance in Favipiravir arm with lesser side effects comparatively. Another randomized clinical trial in China conducted on patients with COVID19 pneumonia (moderate) failed to demonstrate a significant difference in clinical recovery rate at day 7 between Favipiravir (116 patients) versus Umifenovir (112 patients) however, Favipiravir was associated with earlier relief of pyrexia & cough in comparison Another multicenter, open label, randomized phase II/III trial conducted in Russia on moderate COVID19 infection comparing Favipiravir against standard of care in total 60 patients randomized into three treatment groups with 20 patients each: Favipiravir 1600/600 mg, Favipiravir 1800/800 mg, or Standard of care (which included, hydroxychloroquine or chloroquine versus lopinavir/ritonavir versus no etiotropic treatment) concluded that Favipiravir enabled viral clearance in 62.5% patients within 4 days with good safety data, no matter which dosing was used. There has been an observational study on 2141 patients in Japan that showed good recovery among mild (not requiring oxygen), moderate case (requiring oxygen) or younger patients (59 years or younger) whereas poor prognosis in severe (requiring mechanical ventilation or ECMO) or older patients (60 years or older). The most common adverse events were hyperuricemia (335 patients; 15.52%) followed by liver injury or liver function test abnormalities (159 patients; 7.37%) in this study. Similarly, the open label randomized , multicenter clinical trial was conducted in 150 patients to evaluate the efficacy and safety of Favipiravir plus standard supportive care ( Favipiravir treatment arm, versus standard supportive care alone ( control arm ) across seven clinical sites in India.

It was evaluated among mild to moderate patients, randomized within a 48 hours window of testing RT-PCR positive for COVID-19 . The patients received Favipiravir tables of 3,600 mg (1,800 mg BID) (Day 1) + 1,600 mg (800 mg BID) (Day 2 or later) for up to maximum of 14 days , along with standard supportive care . The results from this Phase 3 trial conducted by Glenmark showed numerical improvement for the primary efficacy endpoint with 28.6% faster viral clearance in the overall population (Hazard Ratio 1.367 [95%CI 0.944,1.979]; p=0.129). Additionally , 69.8 % of patients in the Favipiravir treatment arm achieved clinical cure by Day 4, which was statistically significant compared to 44.9% observed in the control group (p=0.019). Likewise, Glenmark's Favipiravir was well tolerated with no serious adverse events or death in the Favipiravir treated arm but adverse events were reported in 26 patients in Favipiravir treatment arm. However, adverse events were mild to moderate and none led to drug discontinuation and dosing adjustments. This trial demonstrated statistically significant faster time to clinical improvement with Favipiravir treatment in Mild to moderate COVID-19 patients compared to the control group. Additionally, An open-label, nonrandomized, before-after controlled study was conducted in an isolation ward of the national clinical research center for infectious diseases at Shenzhen, China.35 patients was enrolled in the FPV arm and the 45 patients in the control arm, all baseline characteristics were comparable between the two arms. From 30 January to 14 February 2020, laboratory-confirmed patients with COVID-19 were consecutively screened, and eligible patients were included in the FPV arm of the study. Patients who had initially been treated with antiviral therapy with LPV/RTV from 24 January to 30 January 2020 were screened, and eligible patients were included in the control arm of the study. The dose was 1600 mg twice daily on Day 1 and 600 mg twice daily on Days 2-14. LPV/RTV (AbbVie Inc., 200 mg/50 mg per tablet) were given orally. The dose was LPV 400 mg/RTV 100 mg twice daily. Both FPV and LPV/RTV were continued until the viral clearance was confirmed or until 14 d had passed. For the 35 patients enrolled in the FPV arm and the 45 patients in the control arm, all baseline characteristics were comparable between the two arms. A shorter viral clearance time was found for the FPV arm versus the control arm (median (interquartile range, IQR), 4 (2.5-9) d versus 11 (8-13) d, P < 0.001). The FPV arm also showed significant improvement in chest imaging compared with the control arm, with an improvement rate of 91.43% versus 62.22% (P = 0.004). After adjustment for potential confounders, the FPV arm also showed a significantly higher improvement rate in chest imaging. Multivariable Cox regression showed that FPV was independently associated with faster viral clearance. In addition, fewer adverse events were found in the FPV arm than in the control arm.In this open-label before-after controlled study, FPV showed better therapeutic responses on COVID-19 in terms of disease progression and viral clearance.These preliminary clinical results provide useful information of treatments for SARS-CoV-2 infection. Doses of Favipiravir ranged widely across studies, from 400 mg up to 6000 mg loading doses, with the more common regimens being 1200 mg per day, split into twice or three times daily doses. 494 Studies were screened, 55 studies assessed for full text eligibility, 29 studies were included. Hyperuricemia was shown as the side effects.

ELIGIBILITY:
A. Inclusion Criteria:

1. Minimum 18 - 80 years of age
2. Clinical Diagnosis of COVID 19 with RT-PCR test for SARS-CoV-2 (If a patient is COVID19 positive based on Antigen test, they can participate in the trial while awaiting result form PCR test with Ct-value)
3. Signed informed consent provided by patient's or patient's healthcare proxy.
4. Fulfills enrollment criteria ( within 6 days of symptoms onset)
5. Willing to practice celibacy OR take contraception during the study & within 7 days after treatment
6. Mild clinical condition with at least 3 of these of these symptoms : fever, cough, malaise/headache
7. Moderate clinical condition with at least 3 of these of these symptoms : fever, cough, malaise/headache

B. Exclusion Criteria:

1. Pregnant (female of childbearing age with positive urine pregnancy test) or miscarriage or within 2 weeks after delivery
2. Severe or critical clinical condition as per NMC clinical guideline for COVID19 Chronic liver with ALT/AST increased 5 times higher than the upper limit of normal or with Child Pugh C
3. Creatinine clearance (Cockcroft-Gault Equation) < 30 ml/min or having hemodialysis/peritoneal dialysis
4. Known allergy or hypersensitivity to Favipiravir
5. Gout or history of gout or hyperuricemia two times the upper limit of normal
6. If using Remdesivir, Lopinavir-ritonavir, Hydroxychloroquine or any other antiviral drug with potential effect against SARS-CoV-2 virus
7. Lactating female
8. Asymptomatic COVID-19 cases
9. Mild COVID-19 cases not meeting the inclusion criteria symptoms
10. Moderate COVID-19 cases not meeting the inclusion criteria symptoms

(*All female patients age 18 - 50 years will be screened for pregnancy by urine test & any pregnant patient will be excluded. Also, the patient must be consented to take contraception or practice celibacy during the study period & until 7 days after treatment. Since the expected wash out period of the study drug Favipiravir is 10hrs minimum to 27.5hrs maximum (half life is 2-5.5hrs), it is a safe practice to avoid conception for 1 week after stopping the drug of interest)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 676 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
clinical improvements in mild cases | 5 day
  Mild cases: Time to clinical improvements is defined as recovery in two out of the three common symptoms that includes fever (body temperature more than 99.5 degrees F), cough, and headache/malaise (scored more than 3 in a pain likert scale of 1 to 10).
  Moderate cases: Time to clinical improvement defined as Improvement in at least 2 out 3 selected common symptoms as above as in mild cases PLUS improvement in shortness of breath (*For the assessment of clinical improvement in moderate cases, we did not include imaging findings because radiological changes lag behind clinical improvement by a few weeks.)
clinical improvements in moderate cases | 10 days
  Moderate Case: Efficacy of Favipiravir on clinical improvement among COVID-19 patients with moderate symptoms compared to Remdesivir

SECONDARY OUTCOMES:
Clinical deterioration in mild & moderate cases | up to 14 days
  In case of mild cases :
  progression of the case into moderate or worse category, as per current NMC guideline, verified/validated by site-PI.
  However, following alarming signs & symptoms should be taken into consideration : patient complaining of shortness of breath or difficulty in breathing, Respiratory rate > 30 per minute, chest pain on coughing or deep breathing, cyanosis of lips & fingertips, feeling dizzy, oxygen saturation < 94 % in room air, etc.
  In case of moderate cases :
  progression of the case into severe or worse category, as per current NMC guideline, verified/validated by site-PI.
Radiological improvement in moderate cases | 11 days
  In moderate cases, chest-X Ray will be done at time of enrollment +/- 24 hours, on day 11 +/- 24 hours & on day 17 +/- 24 hours (if day 11th day chest-X Ray is abnormal) or any time as per clinical decision of the on-site PI.
  Lungs involvement based on Chest X-ray will be categorized into 25 % - 100 % based on visual input by the medical team.
28 days mortality in mold & moderate cases | 28 days
  Any mortality of the study participant, from day of enrollment until 28th day, whether attributed to Favipiravir or other treatment
symptomatic improvement or worsening in mild & moderate cases | 28 days
  Besides the symptoms of primary interest (cough, fever, headache/malaise), the rest of the symptoms are also taken into account & followed for improvement vs worsening
compare change in SARS-CoV-2 viral load in nasopharyngeal swab in mild & moderate cases | 6 days
  Nasopharyngeal swab for RT-PCR test to detect SARS-CoV-2 virus will be performed at screening & day 6 +/- 24 hours to compare the change in viral load, measured by change in Ct (Cycle threshold) value.
  Ct value is indirectly proportional to viral load and has been used as a marker in several studies Ct value > 35 correlates with non-cultivable SARS-CoV-2 viruses
Length of stay in hospital beyond 10 days in mild & moderate cases | 28 days
  Length of stay means total number of days spent in hospital (for mild & moderate cases) after day 10 from day of randomization * (*As of current practice, generally patients with mild or moderate COVID-19 infections are discharged as soon as they are clinically stable , while some cases are held at hospitals until 10th day & sent home without PCR in some sites)

CONTACTS AND LOCATIONS:
Locations (2):
- Nepal (2):
  - Armed Police Force Hospital, Kathmandu, Bagmati
  - Charak Memorial Hospital, Pokhara, Gandaki

IPD SHARING:
Plan to Share IPD: No